CLINICAL TRIAL: NCT05354973
Title: ePRO for the Timely Detection of Side Effects in Cancer Patients Undergoing CAR T Immunotherapy: Feasibility Study (CARTePRO)
Brief Title: ePRO for the Timely Detection of Side Effects in Cancer Patients Undergoing CAR T Immunotherapy
Acronym: CARTePRO
Status: Recruiting | Type: Observational
Sponsor: Stiftung Swiss Tumor Institute (Other)
Collaborators: Klinik Hirslanden, Zurich (Other); Palleos Healthcare GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: KEK ZH: 2021-D0077
Record Dates: First submitted 2022-04-25; First posted 2022-05-02 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Patient Reported Outcome Measures; CAR T-Cell Therapy
Keywords: CAR T-Cell Therapy; ePRO; PRO; Patient Reported Outcome Measure; Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CAR T Cell Treatment
  Interventions: Device: Consilium CareTM

INTERVENTIONS:
Device: Consilium CareTM — This is an observational study using the Consilium CareTM smartphone ePRO application.

SUMMARY:
This study is designed as a feasibility study implementing electronic Patient Reported Outcomes (ePRO) in CAR T treatment for hematological malignancies, in order to describe AE reporting. ePRO assessments will be explored for their feasibility to engage in monitoring and management of CAR T-related toxicities as well as using these digital ePRO tools may improve both, its safety and accessibility.

ELIGIBILITY:
Inclusion Criteria:

1. Signed ICF
2. Patients > 18 years
3. Patients receiving CAR T cell treatment
4. Personal smartphone with iOS or Android system. The operating system must be updated to one of the two newest main versions.

Exclusion Criteria:

1. Patients, whose compliance to the studies' protocol, e.g. due to mental health problems, physical problems, or the private life situation, can be justifiably doubted.
2. Patients with insufficient knowledge about the use of a smartphone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older receiving CAR T Cell therapy and congnitive ability to utilitze a smartphone.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Response time | 84 day +/- 6 days
  Response time in seconds obtained during trail-making test (ePRO) according to daily administration via consilium careTM app, as a potential indicator for ICANS and other CAR T cell therapy-related adverse events.

SECONDARY OUTCOMES:
Occurrence of CRS-related adverse events (ePRO) | 84 day +/- 6 days
  Occurrence of CRS-related adverse events (ePRO): fever, myalgia, rigors, fatigue, and loss of appetite
Number and severity of adverse events (AE) according to the CTCAE | 84 day +/- 6 days
  Number and severity of adverse events (AE) according to the Common Terminology Criteria for Adverse Events (CTCAE) after 12 weeks (ePRO).
  CTCAE on a 5 point scale: Grade 1 is mild, grade 2 moderate, grade 3 severe, grade 4 life-threatening, and grade 5 corresponds to death. Grade 3 and higher correspond to the WHO definition of serious adverse drug reaction ("serious ADR").
Occurrence and type of therapy-associated unplanned consultations | 84 day +/- 6 days
  Occurrence and type of therapy-associated unplanned consultations. Unplanned consultations are defined as additional consultations outside of planned therapy or control visits at the treatment center or with the investigator, as well as unplanned visits to other physicians or emergency services.
Adherence | 84 day +/- 6 days
  Adherence, measured as percentage of days during intervention with electronically captured consilium careTM app usage
Well-being | 84 day +/- 6 days
  Well-being according to the ECOG Performance Status as daily ePRO before and after CAR T cell reinfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Samaras, PD.Dr.med, Principal Investigator — Klinik für Hämatologie und Onkologie
Locations (1):
- Klinik für Hämatologie und Onkologie, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No